CLINICAL TRIAL: NCT00196248
Title: Out-of Hospital Resuscitation Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Other Study IDs: GE IDE No.N00300
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Ventricular Fibrillation; Asystoly; Resuscitation
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Sudden cardiac arrest is one of the most common causes of death in industrial countries. The main objective of this study is to built up a register of all out-of hospital resuscitation in a defined area. According to this register, it is possible to evaluate for example predictors of survival to improve training and organisation of prehospital resuscitations.

ELIGIBILITY:
Inclusion Criteria:

* out of hospital cardiac arrest

Exclusion Criteria:

* none

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Estner, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany